CLINICAL TRIAL: NCT01372735
Title: Clinical Phase I/II Trial to Investigate Neoadjuvant Intensity-Modulated Short Term Radiation Therapy (5x5 Gy) and Intraoperative Radiation Therapy (15 Gy) in Patients With Primarily Resectable Pancreatic Cancer - NEOPANC
Brief Title: Trial of Neoadjuvant Short Course IMRT Followed by Surgery and IORT for Resectable Pancreatic Cancer
Acronym: NEOPANC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Dr. Falk Roeder, Department of Radiation Oncology, University of Heidelberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOPANC
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatic cancer; intensity-modulated radiation therapy; intraoperative radiation therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: neoadjuvant short course IMRT — neoadjuvant short course intensity-modulated radiotherapy, single dose 5 Gy, total dose 25 Gy (5x5 schedule) to primary tumor and regional lymph nodes
Radiation: IORT — intraoperative radiation therapy during resection, 15 Gy (to 90% isodose) to tumor bed

SUMMARY:
The current standard treatment for patients with primarily resectable pancreatic tumors consists of surgery followed by adjuvant chemotherapy. But even in this prognostic favourable group, long term survival is disappointing because of high local and distant failure rates. Postoperative chemoradiation has shown improved local control and overall survival compared to surgery alone but the value of additional radiation has been questioned in case of adjuvant chemotherapy. However, there remains a strong rationale for the addition of radiation therapy considering the high rates of microscopically incomplete resections after surgery. As postoperative administration of radiation therapy has some general disadvantages, neoadjuvant and intraoperative approaches theoretically offer benefits in terms of dose escalation, reduction of toxicity and patients comfort especially if hypofractionated regimens with highly conformal techniques like intensity-modulated radiation therapy are considered.

Therefore the NEOPANC trial has been designed as a prospective, one armed single center study to investigate a combination of neoadjuvant short course intensity-modulated radiation therapy (5x5 Gy) in combination with surgery and intraoperative radiation therapy (15 Gy) followed by adjuvant chemotherapy according to german treatment guidelines in patients with primarily resectable pancreatic cancer. The primary objectives of the NEOPANC trial are to evaluate the general feasibility of this approach and the local recurrence rate after one year. Secondary endpoints are progression-free survival, overall survival, acute and late toxicity, postoperative morbidity and mortality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* histologically confirmed, primary pancreatic cancer of the pancreatic head
* judged as gross completely resectable
* absence of lymph node metastases at the splenic hilum or along the pancreatic tail
* no evidence of distant metastases
* age > 50 years
* Karnofsky performance score ≥ 70%
* adequate bone marrow function (neutrophils > 2000/µl, platelets > 100000/µl)
* adequate renal function (Creatinine < 1.5 mg/dl)
* adequate liver function

Exclusion Criteria:

* missing written informed consent
* missing histological conformation of pancreatic cancer
* judged as gross incomplete or not resectable
* pancreatic cancer located in the pancreatic corpus or tail
* recurrent pancreatic cancer
* incomplete staging
* presence of lymph node metastases along the pancreatic tail or splenic hilum
* presence of distant metastases
* prior radiation therapy to the upper abdominal region
* neoadjuvant chemotherapy or immunotherapy
* participation in another clinical interventional study
* age ≤ 50 years
* other previous or active malignancy (excluding basal cell carcinoma, carcinoma in situ of the cervix)
* Karnofsky performance score <70%
* inadequate bone marrow function
* inadequate renal or liver function
* any other disease or situation, which generally prohibits the use of major surgery or radiation therapy according to the judgement of a surgeon or radiation oncologist
* inability to participate in regular follow up
* pregnancy, inability or incompliance for adequate contraception
* missing ability to give informed consent
* legal custody

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Local recurrence rate | 1 year

SECONDARY OUTCOMES:
Progression-free Survival | up to 5 years from first day of treatment
Overall Survival | up to 5 years from first day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Falk FF Roeder, MD, Principal Investigator — Department of Radiation Oncology, University Hospital Heidelberg; Peter E Huber, MD, PhD, Principal Investigator — Department of Radiation Oncology, German Cancer Research Center (DKFZ); Jens Werner, MD, Principal Investigator — Department of Surgery, University Hospital of Heidelberg
Locations (3):
- Germany (3):
  - Department of Radiation Oncology, German Cancer Research Center, Heidelberg
  - Department of Radiation Oncology, University Hospital Heidelberg, Heidelberg
  - Department of Surgery, University of Heidelberg, Heidelberg

REFERENCES:
- [Derived] Roeder F, Timke C, Saleh-Ebrahimi L, Schneider L, Hackert T, Hartwig W, Kopp-Schneider A, Hensley FW, Buechler MW, Debus J, Huber PE, Werner J. Clinical phase I/II trial to investigate neoadjuvant intensity-modulated short term radiation therapy (5 x 5 Gy) and intraoperative radiation therapy (15 Gy) in patients with primarily resectable pancreatic cancer - NEOPANC. BMC Cancer. 2012 Mar 23;12:112. doi: 10.1186/1471-2407-12-112. PMID 22443802